## **Protocol WI203720**

A Phase 1b/2, Open-Label, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of PF-06252616 in Ambulatory Participants with LGMD2I

# Statistical Analysis Plan (SAP)

Version: 1.0

Author: Nazila Shahri

**Date**: 7-February-2019

# TABLE OF CONTENTS

| 1. AMENDMENTS FROM PREVIOUS VERSION(S) | 7 |
|------------------------------------------------|----|
| 2. INTRODUCTION | 7 |
| 2.1. Study Design | 7 |
| 2.2. Safety Monitoring and Dose Escalation | 8 |
| 2.2.1. Dose Escalation and Stopping Rules | 9 |
| 2.2.2. Safety Monitoring Committee (SMC) | 9 |
| 3. BLINDING | 10 |
| 4. STUDY OBJECTIVES | 10 |
| 4.1. Objectives | 10 |
| 4.1.1. Primary | 10 |
| 4.1.2. Secondary | 10 |
| 4.1.3. Exploratory | 11 |
| 4.2. Endpoints | 11 |
| 4.2.1. Primary Safety | 11 |
| 4.2.2. Secondary Endpoints | 11 |
| 4.2.2.1. Pharmacokinetic | 11 |
| 4.2.2.2. Pharmacodynamic | 11 |
| 4.2.2.3. Strength and Function | 11 |
| 4.2.2.4. Patient Reported Outcomes | 12 |
| 4.2.2.5. Immunogenicity | 12 |
| 4.2.3. Exploratory Endpoint | 12 |
| 4.2.3.1. Pharmacologic | 12 |
| 4.2.3.2. Function | 12 |
| 5. ANALYSIS SETS | 12 |
| 5.1. Full Analysis Set | 12 |
| 5.2. Safety Analysis Set | 12 |
| 5.3. Other Analysis Sets | 12 |
| 5.3.1. PK Concentration Analysis Set | 12 |
| 5.3.2. GDF-8 Concentration Analysis Set | 13 |
| 6. ENDPOINTS AND COVARIATES | 13 |
| 6.1. Safety Endpoints | 13 |
| 6.1.1. Vitals, ECGs and Cardiac Echocardiogram | 13 |

| 6.1.2. Laboratory Data | 13 |
|------------------------------------------------------------------|----|
| 6.1.3. Adverse Events | 14 |
| 6.1.4. Physical Examination/Nose and Throat Exam | 14 |
| 6.2. Secondary Endpoints | 14 |
| 6.2.1. Patient Reported Outcomes | 15 |
| 6.2.2. PK Endpoints | 16 |
| 6.2.3. PD Endpoints | 16 |
| 6.2.4. Columbia-Suicide Severity Rating Scale (C-SSRS) | 16 |
| 6.3. Covariates | 17 |
| 7. HANDLING OF MISSING VALUES | 17 |
| 8. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 17 |
| 8.1. Statistical Methods | 19 |
| 8.2. Statistical Analyses | 19 |
| 8.2.1. Safety Analysis | 19 |
| 8.2.1.1. Adverse Events | 19 |
| 8.2.1.2. Vital Signs | 19 |
| 8.2.1.3. Electrocardiogram | 20 |
| 8.2.1.4. Cardiac MRI/Echocardiogram | 20 |
| 8.2.1.5. Liver MRI | 20 |
| 8.2.1.6. Other Safety Data | 20 |
| 8.2.1.7. Immunogenicity | 20 |
| 8.2.2. Secondary Analyses | 21 |
| 8.2.3. PK Analyses | 22 |
| 8.2.3.1. Concentrations below the limit of quantification | 22 |
| 8.2.3.2. Deviations, missing concentrations and anomalous values | 22 |
| 8.2.3.3. Pharmacokinetic parameters | 22 |
| 8.2.3.4. PK Concentrations | 23 |
| 8.2.4. GDF-8 Analysis | 23 |
| 8.2.4.1. Deviations, missing concentrations and anomalous values | 23 |
| 8.2.4.2. GDF-8 Concentration | 24 |
| 8.2.5. Other Analyses | 24 |
| 8.2.5.1. Exploratory Analyses | 24 |
| 9. REFERENCES | 25 |

| Protocol WI203720 | Statistical Analysis Plan |
|-------------------|---------------------------|
| APPENDIX 1 | |

# LIST OF ABBREVIATIONS

| This is a list of abbrevi | ations that may be used in the SAP. |
|---|---|
| Abbreviation | Term |
| 2MWT | two minute walk test |
| 4SC | four stair climb |
| 10MR | ten meter run |
| ADA | anti-drug antibodies |
| AE | adverse event |
| ALT | alanine transaminase |
| aPTT | activated partial thromboplastin time |
| AST | aspartate transaminase |
| CL | clearance |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DXA | dual energy x-ray absorptiometry |
| ECG | Electrocardiogram |
| FAS | full analysis set |
| FEV1 | Forced expiratory volume in 1 second |
| FSH | follicle stimulating hormone |
| FVC | forced vital capacity |
| GDF-8 | growth differentiation factor 8 |
| GGT | gamma-glutamyl transferase |
| GLDH | glutamate dehydrogenase |
| InQoL | Individualized Neuromuscular Disease Quality of Life |
| IRB | institutional review board |
| IV | intravenous |
| LH | luteinizing hormone |
| LGMD2I | limb girdle muscular dystrophy 2I |
| LVEF | left ventricular ejection fraction |
| LVESV | left ventricular end systolic volume |
| MEP | mean expiratory pressure |
| MIP | mean inspiratory pressure |
| MMT | manual muscle testing |
| MRC | Medical Research Council |
| MRI | magnetic resonance imaging |
| Nab | neutralizing antibodies |
| PK/PD | pharmacokinetic/pharmacodynamics |
| PT | prothrombin time |
| PUL | Performance of Upper Limb |
| RNA | ribonucleic acid |
| SAP | statistical analysis plan |
| SF-36 | Short Form 36 Health Survey |
| SMC | Safety Monitoring Committee |
| SOP | standard operating procedure |
| TEAEs | treatment emergent AEs |

| TIBC | total iron binding capacity |
|------|-----------------------------|
| TUG | timed up and go |

#### 1. AMENDMENTS FROM PREVIOUS VERSION(S)

This is the initial version of the statistical analysis plan.

#### 2. INTRODUCTION

Note: in this document any text taken directly from the protocol is *italicized*.

## 2.1. Study Design

This is a Phase 1b/2, open-label multiple ascending dose study to evaluate the safety, tolerability, efficacy, PK and PD of PF-06252616 administered to in ambulatory participants diagnosed with LGM2I. Three IV infused dose levels administered every 28 days will be investigated in a dose escalating fashion.

*PF-06252616 dose levels:* 

- 5 mg/kg.
- 20 mg/kg.
- 40 mg/kg.

Approximately 20 eligible subjects will be consecutively assigned to 1 of 3 cohorts for approximately 96 weeks (cohort 1) or 64 weeks (cohorts 2 and 3).

## *Cohort 1 (n=4):*

- Lead-in period (16 weeks)
- Treatment A: PF-06252616 5 mg/kg (32 weeks)
- Treatment B: PF-06252616 40 mg/kg (32 weeks)
- Follow-up period (16 weeks)

## *Cohort 2 (n=8):*

- Lead-in period (16 weeks)
- Treatment: PF-06252616 20 mg/kg (32 weeks)
- Follow-up period (16 weeks)

## *Cohort 3 (n=8):*

• Lead-in period (16 weeks)

- Treatment: PF-06252616 40 mg/kg (32 weeks)
- Follow-up period (16 weeks)

At each dose level, subjects will be followed for an initial 16-week lead-in period to establish individual change in disease progression.

The study will begin with 4 subjects being enrolled into Cohort 1. Following the lead-in period, subjects in Cohort 1 will be dosed with 5 mg/kg for a total of 32 weeks (8 doses). Cohort 2 will begin dosing at the mid dose level (20 mg/kg) once safety has been confirmed with subjects in Cohort 1 who have been treated for 16 weeks. Cohort 1 and 3 will begin dosing at the highest dose level (40 mg/kg) once safety has been confirmed with subjects in Cohort 2 who have been treated for 16 weeks.

Each dose level will be evaluated for 32 weeks (8 doses each). Cohort 1 is the only cohort who will receive 2 dose levels (5 mg/kg and 40 mg/kg) and their total treatment time will be 64 weeks.

At the conclusion of the treatment period, subjects will be followed for an additional 16 weeks to monitor for safety, PK and duration of response.



#### 2.2. Safety Monitoring and Dose Escalation

Safety monitoring will be conducted by the Investigator, Pfizer Medical Monitor and an External Medical Monitor. This group will be refered to as the Safety Monitoring Committee (SMC). Safety monitoring by these individuals will include the following reviews:

Dose escalation

- Quarterly safety and
- Ad hoc safety

At each review, a consideration will be made of the number of subjects who have severe AEs or serious AEs in the same organ system which are determined to be related to investigational product. The first dose escalation decision, whether or not to increase from 5 mg/kg in Cohort 1 to 20 mg/kg in Cohort 2 will occur after review of all safety data after the 4<sup>th</sup> subject of Cohort 1 has completed the planned 16 weeks (day 85) or 4 doses. The second dose escalation decision, whether or not to increase from 20 mg/kg in Cohort 2 to 40 mg/kg in Cohorts 1 and 3 will occur after the 4<sup>th</sup> subject in Cohort 2 had completed the planned 16 weeks (day 85) or 4 doses. The SMC may determine it is necessary to close or adjust a dose level within the study.

### 2.2.1. Dose Escalation and Stopping Rules

Table 1. Criteria to Determine Dose Escalation or Stopping

| DECISION | CRITERIA |
|---|---|
| Dose Escalation | SMC review of aggregate safety data from either: |
| | • Cohort 1 (n=4) 16 weeks (day 85) <u>or</u> |
| | • Cohort 2 (n=4) 16 weeks (day 85) |
| | and agree that safety is met <u>and</u> |
| | The estimate as determined by R2* value is within the normal range (R2* $\leq$ 139 Hz at 3.0 T) $^{1,2,3}$ |
| No Escalation, Stop | SMC review of aggregate safety data from either: |
| Dosing | • Cohort 1 (n=4) 16 weeks (day 85) <u>or</u> |
| | • Cohort 2 (n=4) 16 weeks (day 85) |
| | And agree that the current dose is not safe or |
| | The liver iron content estimate as determined by $R2^*$ value is above the "mild overload" range for any subject within the cohort ( $R2^* > 369$ Hz at 3.0 T) $^{1,2,3}$ |

If dosing is terminated at any dose level, subjects will continue to be followed for resolution of the safety finding or until a new baseline is established. Depending on the nature of the reason for stopping dosing, the SMC will consider if the enrolled subjects can be continued at a lower dose level.

#### 2.2.2. Safety Monitoring Committee (SMC)

The SMC will be composed of three members: The Investigator, Pfizer Medical Monitor and an External Medical Monitor. The External Medical Monitor will be a clinical trialist and an expert in the neuromuscular field. The External Medical Monitor will not be a member of the Investigator's institutions (Johns Hopkins School of Medicine [JHSOM] and Kennedy Krieger Institute [KKI]) nor an employee of Pfizer. The SMC will be responsible for ongoing safety monitoring from the initiation of the study through the final study visit. Reviews will

include aggregate safety, targeted medical events of special interest including liver toxicity, and serious AE data. The SMC may also complete ad hoc safety reviews. Ad hoc PK data may be provided to the SMC as requested.

Following the data review, the SMC will determine if the study should be continued with no changes, modified, or stopped (eg, due to safety). Decision to continue the study must be unanimous. Decision to stop the study can be made by any of the three members. In all other decisions, the External Medical Monitor will cast the deciding vote. The recommendations made by the SMC to modify the study will be forwarded to JHSOM IRB for final decision. At any time the SMC may indicate that the limit of safety and/or tolerability has been reached and that any of the dose levels will be removed from the study.

The SMC will consider the following safety criteria during their safety review:

- The number of subjects who have severe AEs or serious AEs in the same organ system which are determined to be related to study medication.
- Other findings that indicate that dose escalation should be halted.

#### 3. BLINDING

This study is open label. Subjects, investigators and pharmacists will be aware of the active treatment and dose level.

#### 4. STUDY OBJECTIVES

## 4.1. Objectives

## **4.1.1. Primary**

• To determine the safety and tolerability of multiple ascending repeat IV doses of PF-06252616 in ambulatory participants with LGMD2I.

#### 4.1.2. Secondary

- To assess the PK exposures of PF-06252616 in LGMD21.
- To evaluate the PD activity of PF-06252616 based on the percent change of muscle volume as measured on MRI compared to baseline.
- To evaluate the PD activity of PF-06252616 based on GDF-8 (myostatin) modulation in blood and in tibialis muscle.
- To characterize the functional effects of PF-06252616 on muscle strength and functional assessments compared to baseline.
- To characterize the effects of PF-06252616 on respiratory function compared to baseline.

- To characterize the effects of PF-06252616 on Patient reported outcome measures.
- To evaluate the immunogenicity of PF-06252616.

## 4.1.3. Exploratory

• To evaluate functional outcome measures in LGMD2I.

## 4.2. Endpoints

## 4.2.1. Primary Safety

- Incidence of dose limiting or intolerability treatment related AEs by day 337 or 561.
- Incidence, severity and causal relationship of treatment emergent AEs (TEAEs) and withdrawals due to TEAEs by day 337 or 561.
- Incidence and magnitude of abnormal laboratory findings (clinical laboratory tests [hematology, chemistry], GGT, GLDH, PT, aPTT, creatine kinase, amylase, serum ferritin, serum iron, % transferrin saturation, Total Iron Binding Capacity (TIBC), LH, FSH, estrogen, cardiac troponin I, fecal occult blood and urinalysis) by day 337 or 561.
- Abnormal and clinically relevant changes in liver MRI and physical examinations, weight, vital signs, ECG, echocardiogram measured LVEF, DXA (bone mineral density), menstruation cycle as monitored by diary and C-SSRS (See Appendix 1 And Appendix 2 of the protocol) parameters by day 337 or 561.

## 4.2.2. Secondary Endpoints

#### 4.2.2.1. Pharmacokinetic

• All subjects receiving active drug: serum PF-06252616  $C_{max}$  and  $C_{trough}$  for all visits with PK collections and at steady-state.

#### 4.2.2.2. Pharmacodynamic

- Mean percent change from baseline in muscle volume as measured on MRI.
- Total serum GDF-8 concentrations for all visits with GDF-8 collections

#### 4.2.2.3. Strength and Function

- Mean change from baseline on function tests including PUL, Timed up-and-go (TUG), 10-meter walk/run (10MR), 2-meter walk test (2MWT), and 4 stair climb (4SC).
- Mean change from baseline on pulmonary function tests including forced vital capacity (FVC), FEV1(forced expiratory volume in 1 second), maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).

• Mean change from baseline on muscle strength by manual muscle test (MMT) and Hand-Held dynamometry.

## **4.2.2.4. Patient Reported Outcomes**

• Mean change from baseline on Patient reported outcomes (InQoL, SF-36)(See Appendix 3 and Appendix 4 of the protocol).

## 4.2.2.5. Immunogenicity

• Incidence of ADA and NAb development.

## 4.2.3. Exploratory Endpoint

## 4.2.3.1. Pharmacologic

- *Mean percent change from baseline in lean body mass by DXA.*
- Mean percent change from baseline in muscle quality (fat infiltration) as measured by quantitative Dixon.
- Mean change from baseline in muscle quality as measured by T1/STIR.

#### **4.2.3.2. Function**

• Evaluate the utility and changes from baseline of Functional Workspace as an outcome measure for LGMD2I.

### 5. ANALYSIS SETS

#### 5.1. Full Analysis Set

All analyses will be based on the full analysis set (FAS) which includes all enrolled subjects who have received at least one dose of study drug.

#### 5.2. Safety Analysis Set

Safety analyses will be based on the full analysis set.

## 5.3. Other Analysis Sets

## 5.3.1. PK Concentration Analysis Set

The PK concentration population is defined as all enrolled subjects who received at least 1 dose of PF-06252616 and in whom at least 1 concentration value is reported.

## 5.3.2. GDF-8 Concentration Analysis Set

The GDF-8 concentration population is defined as all enrolled subjects in whom at least 1 concentration value is reported.

#### 6. ENDPOINTS AND COVARIATES

## 6.1. Safety Endpoints

Safety data will be summarized according to current Pfizer data standards including incidence of anti-drug antibodies and neutralizing antibodies by days 1 (to capture low dose safety) and 561 (last visit) for cohort 1 and day 337 (last visit) for cohorts 2 and 3.

At the screening visit, the "Baseline/Screening" assessment from the Columbia Suicide Severity Rating Scale will be performed. At all other visits the "Since Last Visit" assessment will be performed. The score at the screening visit will be the baseline. All adverse events will be reported under the treatment last received prior to the onset of the adverse event.

## 6.1.1. Vitals, ECGs and Cardiac Echocardiogram

Baseline values for vital signs, ECG and Cardiac Echocardiogram will be the last acceptable pre-dose measurement taken either on the day of dosing or at the baseline or screening visit.

If not supplied, QTcF will be derived using Fridericia's heart rate correction formula: QTcF = QT / (RR) $^{(1/3)}$ , where RR = 60/HR (if RR is not provided).

Echocardiograms should be collected at times specified in the Schedule of Activities (please see protocol). To ensure safety of the subjects, a qualified individual at the investigator site will evaluate the echocardiogram for ejection fraction (EF) and left ventricular end systolic volume (LVESV).

## 6.1.2. Laboratory Data

Using the current Pfizer data standards, the last pre-dose value before the first day of dosing is used as the baseline for all laboratory parameters.

Clinical laboratory tests include hematology with complete blood count and differential, comprehensive metabolic panel (sodium, potassium, chloride, carbon dioxide, blood urea nitrogen, creatinine, calcium, glucose, total protein, albumin, total bilirubin, AST, ALT, alkaline phosphatase), cardiac troponin I, gamma-glutamyl transferase (GGT), prothrombin time (PT), activated partial thromboplastin time (aPTT), creatine kinase, amylase and urinalysis. If total bilirubin is abnormal, direct bilirubin will be tested reflexively. The samples for serum ferritin, serum iron, transferrin saturation and TIBC should be collected in the morning following an 8 hour fast. Hormone testing will include LH,FSH and estrogen in female subjects only. Laboratory monitoring will also be performed to detect ADA and NAb.

#### 6.1.3. Adverse Events

Severity is the key baseline information for adverse events. To judge an increase in adverse event severity after dosing, the post-dosing adverse event severity will be compared to the adverse event severity reported prior to the first day of study drug administration will be used.

## 6.1.4. Physical Examination/Nose and Throat Exam

The physical examination will include head,ears,eyes,nose,mouth,skin,heart and lung examinations, lymph nodes, gastrointestinal musculoskeletal, and neurological systems. A targeted and throat muscosal exam will be performed according to the Protocol's Schedule of Activities to monitor for any signs of mucosal telangiectasias.

## **6.2. Secondary Endpoints**

- Mean change from baseline on function tests including PUL, Timed up-and-go (TUG), 10-meter walk/run (10MR), 2-meter walk test (2MWT), and 4 stair climb (4SC).
- Mean change from baseline on pulmonary function tests including forced vital capacity (FVC), FEV1(forced expiratory volume in 1 second), maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).
- Mean change from baseline on muscle strength by manual muscle test (MMT) and Hand-Held dynamometry.

#### **Functional Assessment:**

Functional assessments will be obtained according to the Protocol Schedule of Activities. In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessments will be performed after the MRI and before needle muscle biopsy whenever possible. All functional assessments will be conducted by a trained physiotherapist.

## **Pulmonary Function**

Pulmonary function testing will be completed to evaluate the maximal lung function recording FVC, FEV1, MIP and MEP.

## 4 Stair Climb (4 SC)

The 4 SC quantifies in seconds the time required for a subject to ascend 4 standard steps. The method the subject uses (eg, using the hand rails) to climb the stairs is recorded to understand any change in technique that occurs over time.

#### **Two Minute Walk Test (2MWT)**

The 2-minute walk test (2MWT) is a shorter measure of walking performance than the 6-minute walk test (6MWT). In this test, subjects start from a clearly marked line of tape on the

floor and walk up and down a 21 meter hallway for 2 minutes at a fast but comfortable speed wearing their regular footwear.

#### 10-meter walk/run

The 10-meter walk/run is a frequently used timed function test in muscular dystrophy trials demonstrating good test-retest reliability in several different populations and has been used in studies of LGMD2I <sup>19,27</sup>. Individuals are instructed to walk at a fast but comfortable speed in a long cooridor with an even surface. Measurement of time begins at a still-standing start and stops when the individual passes the 10-meter mark while continuing to walk 2.5 meters beyond the mark.

## Timed Up & Go (TUG)

The Timed Up & Go is a measure of hip strength as well as dynamic balance. This timed function test has good test-retest reliability and has been used in studies of LGMD2I <sup>19,27</sup>. The individual is asked to rise from a seated position in a standardized armchair (44-45 cm), walk at a comfortable and safe pace to a tape mark on the floor 3 meters away, turn around the mark, go back to the chair, turn and sit down.

## **Strength Assessment**

Muscle strength will be quantified by means of manual muscle testing (MMT) quantified by the modified Medical Research Council (MRC) scale and by handheld dynamometer quantified in pounds (lbs). The following muscle groups will be evaluated: shoulder abduction, elbow flexion, elbow extension, hip extension, hip flexion, knee extension, knee flexion.

## Performance of Upper Limb (PUL)

The PUL scale has been devised to assess motor performance of the upper limb. Motor performance will be impacted by muscle strength and contractures and the scale aims to incorporate performance of shoulder, elbow, wrist and hand function.

For all the above endpoints except forced vital capacity, more than one assessment may be performed at the site. If more than one assessment is performed, the site is to record the best (maximum) score in the case report forms. For the forced vital capacity, 3 attempts will be made and the percent predicted will be calculated based on the maximum forced vital capacity.

## **6.2.1. Patient Reported Outcomes**

• Mean change from baseline on Patient reported outcomes (InQoL, SF-36)(See Protocol Appendix 3 and Appendix 4).

#### InQoL

InQoL survey consists of 45 questions within 10 sections. Four sections focus on the impact of key muscle disease symptoms (weakness, locking, pain, and fatigue), five look at the

impact (degree and importance of impact) muscle disease has on particular areas of life, and one section asks about the positive and negative effects of treatment<sup>4</sup>.

#### **SF36**

SF-36 questionnaire is a multi-purpose, short form patient-reported health survey with only 36 questions. It is a generic measure, providing an 8-scale profile of functional health as well as measuring physical and mental health. Each scale is transformed into a 0-100 scale, with a score of 0 being equivalent to maximum disability and a score of 100 being indicative of no disability<sup>5</sup>. It provides a measure of relative disease burden and allows differentiating the health benefits produced by various different treatments.

## 6.2.2. PK Endpoints

Blood samples for PK analysis of PF-0625616 will be taken according to the Schedule of Activities in the protocol. Serum PF-06252616 concentration data for the following subjects and visits will be derived.

• All subjects receiving active drug:  $C_{max}$ , and  $C_{trough}$  for all visits with PF-06252616 dosing.

## 6.2.3. PD Endpoints

The baseline for all pharmacodynamics endpoints is the last pre-dose value before the first day of dosing.

Graphical analysis of total GDF-8 levels as absolute and percentage of baseline will be performed. Analyses will be employed to determine the effects of dose and concentration on the GDF-8 levels over time. The GDF-8 concentrations will be summarized descriptively by treatment and time points.

#### **6.2.4.** Columbia-Suicide Severity Rating Scale (C-SSRS)

The C-SSRS will be evaluated at times specified in the Schedule of Activities of the protocol. The Baseline/Screening (Version 1/14/09) (Appendix 1 of the protocol) of the C-SSRS should be completed at the Screening Visit (Visit 1). At all study visits following the Screening Visit, the Since Last Visit (Version 1/14/09) (Appendix 2 of the protocol) of the C-SSRS should be utilized. The Since Last Visit version refers to the subject's experience since their last visit.

At Screening or Baseline, if the subject endorses a 4 or 5 on the C-SSRS ideation section or reports any suicidality behavior, then the subject is not eligible for study participation and an evaluation of suicide risk (risk assessment) must be completed.

At every visit after Screening, if the subject endorses a 4 or 5 on the C-SSRS ideation section or reports any suicidality behavior, then the subject must be discontinued as outlined in Section 6 of the protocol, Subject Withdrawal and evaluation of suicide risk (risk assessment) must be completed.

#### 6.3. Covariates

Covariates will be summarized for the FAS and by treatment. Continuous baseline covariates will be summarized by: n, mean, median, standard deviation, min and max. Binary and factor covariates will be summarized by percent and counts.

Additional covariates including the qualitative assessment for the 4SC will be summarized over time and may be explored in the modeling of the 4SC statistical analysis.

#### 7. HANDLING OF MISSING VALUES

Missing data for the secondary endpoints will be imputed using maximum likelihood techniques for a mixed effects model. This analysis is unbiased under the assumption of missing at random when the model assumptions hold. Subjects who lose motor functions (e.g. TUG, 2MWT) will be regarded as missing not at random. Additional imputation methods to assess the sensitivity of the analysis to missing not at random data may also be performed. A completer analysis will also be conducted as a sensitivity analysis.

Missing data for the patient reported outcome will be handled according to the guidance of the developers.

Laboratory values below the limit of quantification will be analyzed at the limit of quantification for that parameter except for PK data. For laboratory listings, the <BLQ will be used with the actual limit of quantification used in place of BLQ.

#### 8. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

Continuous variables will be summarized by the number (N), mean, median, standard deviation, minimum and maximum. Categorical variables will be summarized by percent and counts. All summaries will be displayed by treatment. Efficacy data will be listed, tabulated and graphically represented, as appropriate.

All analyses will be based on the full analysis set (FAS) which includes all enrolled subjects who have received at least one dose of study drug.

Below is outlining the definition of baseline for secondary endpoints:

As per Figure 1 below shows each treatment period has been divided into 16 week intervals. Endpoint is the change from the baseline to the subsequent 16<sup>th</sup> week.

A placebo group is constructed by combining the 3 cohort's running periods. Each cohort has an initial 16 week running period, they are combined together to form a placebo group which will be used as a comparison group, testing against active treatments. There will be a total of 20 subjects in the placebo group.

For cohort 1 the first comparison would be: placebo (3 cohort's running periods) vs. active treatment (1<sup>st</sup> interval) which starts from the end of the running period to the end of the first 16 weeks of active treatment i.e. week 17 to week 32. The next comparison would be placebo

vs. active treatment (second interval) which starts from the end of the second 16 week active treatment i.e. week 33 to week 48. Then the next comparison would be placebo vs. active treatment (third interval) i.e. week 49 to week 64. Finally comparing placebo vs. active treatment (fourth interval) i.e. week 65 to week 80, as shown in the table 1 below.

The above rational is to be used for cohorts 2 and 3.

To conclude there will be 8 statistical tests.

Table 1. Active Treatment Intervals

| Active treatment Intervals | | |
|----------------------------|----------|----------|
| Cohort 1 | Cohort 2 | Cohort 3 |
| 17-32 | 17-32 | 17-32 |
| 33-48 | 33-48 | 33-48 |
| 49-64 | | |
| 65-80 | | |

Figure 1. LGMD2i Active vs. "Placebo" 16 weeks 32 weeks 32 weeks 16 weeks Follow-Lead-In Cohort 1 N=4 up Baseline of Baseline of Baseline of Baseline Baseline of Active Active Placebo Follow-Cohort 2 N=8 Lead-In up Baseline of Active Follow-Cohort 3 N=8 Lead-In up Baseline of Active

#### 8.1. Statistical Methods

The planned statistical methods and analyses for the primary and all secondary endpoints are described in detail in Section 8.2.1 and Section 8.2.2 below.

To explore the data further and to assess the goodness-of-fit of all statistical models, separate SAS datasets will be provided by the clinical programmer to the statistician. Covariates for data exploration may include baseline and/or demographic covariates such as gender, age, weight (continuous and/or Pfizer standard categorical cut-offs), site, country, etc.

## 8.2. Statistical Analyses

Subject evaluation groups will show end of study subject disposition and will show which subjects were analyzed for safety (adverse events and laboratory data), pharmacokinetics (PK) and all secondary efficacy measures (FAS). Frequency counts will be supplied for subject discontinuation(s) by treatment. Data will be reported in accordance with the sponsor reporting standards.

A breakdown of demographic data will be provided for age, race, weight, body mass index, and height. Each will be summarized by treatment cohort in accordance with the sponsor reporting standards.

The following data will also be summarized by treatment and in accordance with the current sponsor reporting standards:

Discontinuations, adverse events, laboratory data, vital signs, ECG and concomitant medication data will be summarized by treatment and in accordance with current Pfizer data standards.

#### 8.2.1. Safety Analysis

For all safety variables and vital signs, the baseline will be predose measurement taken either on the day of dosing or at the baseline or screening visit.

#### 8.2.1.1. Adverse Events

All adverse event summaries will be presented for the complete study. Additionally, summary tables of the most frequent adverse events will be presented by cohorts. Based on the review of the frequency and timing of adverse events, additional summaries may be requested.

## **8.2.1.2.** Vital Signs

Systolic blood pressure, diastolic blood pressure and pulse rate will be listed and tabulated by dose group and week with descriptive statistics. Change from baseline will also be summarized using the same descriptive statistics by dose group and visit.

## 8.2.1.3. Electrocardiogram

The following ECG data will be listed: QT, QTc (Fridericia's), heart rate, QRS duration, PR and RR interval.

Baseline and change from baseline for QT, QTcF, heart rate, QRS, PR and RR will be summarized using descriptive statistics by treatment and study week. Any triplicate measurements will be averaged prior to the calculation of summary statistics. For QTcF a classification of absolute values and increase from baseline will be used.

The number of subjects with average of the triplicate QTcF < 450 ms,  $450 \text{ ms} \leq QTcF < 480 \text{ ms}$ ,  $480 \text{ ms} \leq QTcF < 500 \text{ ms}$  and QTcF values  $\geq 500 \text{ ms}$  will be tabulated by treatment and visit. The number of subjects with maximum increase from baseline QTcF < 30 ms,  $30 \text{ ms} \leq QTcF < 60 \text{ ms}$  and  $QTcF \geq 60 \text{ ms}$  will be tabulated by treatment and study week. In addition, the number of subjects with uncorrected QT values  $\geq 500 \text{ ms}$  will be summarized.

Triplicate measures will be averaged prior to categorizing subjects. However, the number of subjects with any single uncorrected QT value  $\geq$ 500 ms (not the average) will be summarized.

#### 8.2.1.4. Cardiac MRI/Echocardiogram

The mean absolute and percent change from baseline in LVEF and LVESV will be evaluated. LVEF shift tables will be prepared for cohorts and the total.

#### 8.2.1.5. Liver MRI

The mean absolute and percent change from baseline in the R2\* value will be tabulated for each subject. Summaries of the categorical assessment of iron overload (normal, above normal, etc.) will be presented.

## 8.2.1.6. Other Safety Data

C-SSRs, DXA (spine and hip), prior medication(s), medical history and physical examination will be listed in accordance with the sponsor reporting standards but not subjected to formal statistical analysis.

Any other screening data that is captured on the study database will be listed.

#### 8.2.1.7. Immunogenicity

Immunogenicity analysis will be based on the immunogenicity analysis population which will be the same as the safety analysis population. This will include anti-drug antibody and neutralizing antibody development by all visits with ADA samples until the end of follow-up. Both continuous endpoints (titer) and categorical endpoints (i.e. positive, negative and inconclusive) will be reported for the anti-drug antibody and neutralizing antibody assays by dose and sampling time points. Data permitting, the incidence of anti-drug antibody and neutralizing antibody will be summarized by time points within each dose cohort and may be

also summarized by dose. The impact of anti-drug antibody and neutralizing antibody on PK and PD parameters and profiles, efficacy and safety may be also evaluated but no formal statistical inference will be drawn.

## 8.2.2. Secondary Analyses

The secondary endpoints, change from baseline in FVC, muscle strength, timed function tests and patient reported outcome measures, will be analyzed based on the FAS using a mixed effects model with REML estimation. The change over the lead-in period, treatment, time and treatment by time interaction and will be included as fixed effects in the model. The following covariance structures and random effects will be considered: Marginal Unstructured, Marginal Variance Components, Marginal Compound Symmetry, Variance Components with Random Intercept, Unstructured with Random Intercept and Slope, Compound Symmetry with Random Intercept and Slope, Spatial Linear with Random Intercept and Slope. Choice of final model will be based on minimum AIC.

.

The dependent variable: change from Visit 3 at each *post-baseline interval*, i.e.:

Change over post-baseline interval 1: (visit 7 –visit 3)

Change over post-baseline interval 2: (visit 11-visit 3)

Change over post-baseline interval 3: (Visit 15-Visit 3), for Cohort 1 only

Change post-baseline interval 4: (Visit 19-Visit 3), for Cohort 1 only

#### Covariates are:

- Fixed effects:
  - o Baseline interval change (Visit 3 Visit 2)
  - O Treatment category (Dose= "5mg/kg", "5 + 40 mg/kg", "20mg/kg" or "40mg/kg")
  - o Time coded as Interval Indicator
  - o Treatment category by time interaction
- Random effects:
  - Choice among Marginal Model, Random Intercept Model, and Random Intercept and Slope are selected based on the minimum AIC

Model-estimated change over each post-baseline interval with, 95% two-sided confidence intervals, will be displayed in tabular format.

For each dose level graphical displays will show model-based estimates of change in the mean functional measure from visit 3 at each visit and corresponding confidence intervals derived from the model.

Additionally a completer analysis will also be conducted as a sensitivity analysis for the missing data handling under the mixed effects modeling. The completer analysis will only

include subjects that completed all assessments at the last scheduled visit using the same longitudinal mixed effects model as the primary analysis.

*Transformation of the data will be considered if model assumptions are not met.* 

## 8.2.3. PK Analyses

## 8.2.3.1. Concentrations below the limit of quantification

In all data presentations (except listings), concentrations below the limit of quantification (BLQ) will be set to zero. (In listings BLQ values will be reported as "<LLQ", where LLQ will be replaced with the value for the lower limit of quantification.)

#### 8.2.3.2. Deviations, missing concentrations and anomalous values

In summary tables and plots of the median values at each time point, statistics will be calculated having set concentrations to missing if 1 of the following cases is true:

- 1. A concentration has been collected as ND (i.e. not done) or NS (i.e. no sample),
- 2. A deviation in sampling time is of sufficient concern or a concentration has been flagged anomalous by the pharmacokineticist.

Note that summary statistics will not be presented at a particular time point if more than 50% of the data are missing.

#### 8.2.3.3. Pharmacokinetic parameters

Nominal PK sampling times will be used in the derivation of PK parameters.

If a PK parameter cannot be derived from a subject's concentration data, the parameter will be coded as NC (i.e. not calculated). (Note that NC values will not be generated beyond the day that a subject discontinues.)

In summary tables, statistics will be calculated by setting NC values to missing; and statistics will not be presented for a particular treatment if more than 50% of the data are NC. For statistical analyses (i.e. analysis of variance), PK parameters coded as NC will also be set to missing.

If an individual subject has a known biased estimate of a PK parameter (due for example to an unexpected event such as incomplete administration of the IV infusion dose), this will be footnoted in summary tables and will not be included in the calculation of summary statistics.

The PK parameters will be listed and summarized for subjects in the PK parameter analysis set. Parameters will be summarized by cohort and dose. Each PK parameter will include the set of summary statistics as specified in the table below:

#### Table 3. PK Parameters

| Parameter | Summary Statistics |
|---|---|
| Cmax, Ctrough, | N, arithmetic mean, median, cv%, standard deviation, minimum, maximum, geometric mean, geometric CV% |

#### 8.2.3.4. PK Concentrations

To assess the PK profile of PF-06252616, PK concentrations will be listed, summarized and plotted for subjects in the PK analysis set, where missing and BLQ values will be handled as detailed in Section 8.2.4.2.

Presentations for PF-06252616 will include:

- A listing of all concentrations sorted by dose, subject ID, cohort and nominal time postdose. The listing of concentrations will include the actual sample collection times, and the time of dosing. Deviations from the nominal time will be given in a separate listing.
- A summary of concentrations by cohort, dose and nominal time postdose, where the set of statistics will include n, mean, median, standard deviation, coefficient of variation (cv), minimum, maximum and the number of concentrations above the lower limit of quantification.
- Median trough (predose) concentrations against nominal dosing week by cohort and dose. Individual subject trough concentrations will also be plotted. Linear scale.
- Median concentrations at the end of infusion (nominally at 2 hour post start of infusion)
  against nominal dosing week by cohort and dose, as described above for trough
  concentrations. Individual subject end of infusion concentrations will also be plotted.
  Linear scale.

The range for the x-axes of these plots will be decided on review of the data, and will depend on how long PF-06252616 concentration is quantifiable in the matrix.

For summary statistics and median plots by sampling time, the nominal PK sampling time will be used. For individual subject plots by time, the actual PK sampling time will be used.

## 8.2.4. GDF-8 Analysis

#### 8.2.4.1. Deviations, missing concentrations and anomalous values

In summary tables and plots of the median values at each time point, statistics will be calculated having set concentrations to missing if 1 of the following cases is true:

1. A concentration has been collected as ND (i.e. not done) or NS (i.e. no sample),

2. A deviation in sampling time is of sufficient concern or a concentration has been flagged anomalous by the pharmacokineticist.

Note that summary statistics will not be presented at a particular time point if more than 50% of the data are missing.

#### 8.2.4.2. GDF-8 Concentration

To assess the PD profile of PF-06252616, GDF-8 concentrations will be listed, summarized and plotted for subjects in the PD analysis set, where missing the data will be handles as outlined in Section 8.2.5.1.

- A listing of all concentrations sorted by dose, subject ID, cohort and nominal time postdose. The listing of concentrations will include the actual sample collection times, and the time of dosing. Deviations from the nominal time will be given in a separate listing.
- A summary of concentrations by dose, cohort and nominal time postdose, where the set
  of statistics will include n, mean, median, standard deviation, coefficient of variation
  (cv), minimum, maximum and the number of concentrations above the lower limit of
  quantification.
- Median total GDF-8 concentrations and Change from Baseline against nominal time postdose by cohort and Dose. Linear scale.
- Mean total GDF-8 concentrations and Change from Baseline against nominal time postdose by cohort and Dose. Linear scale.
- Individual total GDF-8 concentrations and Change from Baseline against actual time postdose by cohort and Dose (including all subjects). Linear scale.

The range for the x-axes of these plots will be decided on review of the data, and will depend on how long GDF-8 concentration is quantifiable in the matrix.

For summary statistics and median plots by sampling time, the nominal GDF-8 sampling time will be used. For individual subject plots by time, the actual GDF-8 sampling time will be used.

#### 8.2.5. Other Analyses

## 8.2.5.1. Exploratory Analyses

All exploratory endpoints, including the pharmacologic and health outcome endpoints will be summarized by treatment group. Additional analyses may be performed to understand the relationship between these endpoints and treatment.

*Any population PK/PD analysis conducted will be reported separately.* 

Additionally, data permitting, relationships between PF-06252616 PK, GDF-8, imaging data (DXA, MRI), functional assessment, immunogenicity and any safety signals may be explored.

#### 9. REFERENCES

- Hankins, J. S. et al. R2\* magnetic resonance imaging of the liver in patients with iron overload. Vol. 113 (2009).
- Wood, J. C. et al. MRI R2 and R2\* mapping accurately estimates hepatic iron concentration in transfusion-dependent thalassemia and sickle cell disease patients. Vol. 106 (2005).
- Storey, P. *et al.* R2\* imaging of transfusional iron burden at 3T and comparison with 1.5T. *Journal of Magnetic Resonance Imaging* **25**, 540-547, doi:10.1002/jmri.20816 (2007).
- 4 Marshall, W. A. & Tanner, J. M. Variations in the Pattern of Pubertal Changes in Boys. *Arch Dis Child* **45**, 13-23 (1970).
- Ware, J. E. SF-36 Health Survey Update. *Spine* **25**, 3130-3139 (2000).

# APPENDIX 1.

# **Planned Data Display**

| Item | Number | Title Population | |
|---|---|---|---|
| | | ENROLLMENT AND DISPOSITION | |
| Table | Table 14.1.1.1 | Subject Evaluation Groups by Cohort | All Enrolled Subjects |
| Listing | Table 14.1.1.2 | Subject Evaluation Groups | All Enrolled Subjects |
| Listing | Table 14.1.1.3 | Subject Discontinuation | All Enrolled Subjects |
| | | DEMOGRAPHICS | |
| Table | Table 14.1.1.4 | Subject Demographics and Baseline Characteristics | FAS |
| Listing | Table 14.1.1.5 | Subject Demographics and Baseline Characteristics | FAS |
| Listing | Table 14.1.1.6 | Clinical Significance of Physical Examination | FAS |
| | | Study Drug | |
| Table | Table 14.1.1.7 | Summary of Number of Subjects by Cohort and Dose Level | FAS |
| Listing | Table 14.1.1.8 | Administration Schedule | FAS |
| Listing | Table 14.1.1.9 | Infusion Site Assessment | FAS |
| Listing | Table 14.1.1.10 | Dose Administration by Dose Level and Visit | FAS |
| Listing | Table 14.1.1.11 | Dose Administration by Dose Level, Cohort and Visit | FAS |
| Listing | Table 14.1.1.12 | Dose Administration by Cohort, Total and Visit | FAS |
| | | Safety | |
| Table | | Treatment-Emergent Adverse Events (All Causalities) by | FAS |
| | Table 14.1.1.13 | Dose Level and Cohort | |
| Table | | Treatment-Emergent Adverse Events (All Causalities) by | FAS |
| | Table 14.1.1.14 | Cohort and Total | |
| Table | | Incidence and Severity of Treatment-Emergent Adverse | FAS |
| | Table 14.1.1.15 | Events by Dose Level and Cohort (All Causalities) | |
| Table | | Incidence and Severity of Treatment-Emergent Adverse | FAS |
| | Table 14.1.1.16 | Events by Cohort and Total (All Causalities) | |
| Table | m 11 11 1 1 1 1 5 | Treatment-Emergent Adverse Events (Treatment Related) by | FAS |
| TD 11 | Table 14.1.1.17 | Dose Level and Cohort | E+C |
| Table | T 11 14 1 1 10 | Treatment-Emergent Adverse Events (Treatment Related) by | FAS |
| Tabla | Table 14.1.1.18 | Cohort and Total | EAC |
| Table | Table 14.1.1.19 | Incidence and Severity of Treatment-Emergent Adverse | FAS |
| Table | 1 abie 14.1.1.19 | Events by Dose Level and Cohort (Treatment Related) Incidence and Severity of Treatment-Emergent Adverse | FAS |
| Table | Table 14.1.1.20 | Events by Cohort and Total (Treatment Related) | TAS |
| Table | 14010 14.1.1.20 | Serious Adverse Events by System Organ Class by Dose | FAS |
| Table | Table 14.1.1.21 | Level and Cohort (All Causalities) | TAS |
| Table | 14010 1 1.11.121 | Serious Adverse Events by System Organ Class by Cohort | FAS |
| 1 40010 | Table 14.1.1.22 | and Total (All Causalities) | |
| Table | | Serious Adverse Events by System Organ Class by Dose | FAS |
| | Table 14.1.1.23 | Level and Cohort (Treatment Related) | |
| Listing | Table 14.1.1.24 | Discontinuations Due to Adverse Events | FAS |
| Listing | Table 14.1.1.25 | Adverse Events | FAS |
| Listing | Table 14.1.1.26 | Individual Listing of Deaths | FAS |
| Listing | Table 14.1.1.27 | Serious Adverse Events | FAS |
| Listing | Table 14.1.1.28 | Treatment Related Serious Adverse Events | FAS |
| | | Clinical Laboratory | |
| Table | | Incidence of Laboratory Test Abnormalities (without Regard | FAS |
| | Table 14.1.1.29 | to Baseline Abnormality) by Dose Level and Cohort | |
| Table | Table 14.1.1.30 | Serum Iron Indices (Total Iron Binding Capacity, Serum Iron, | FAS |
| | | | 1 |

| _ | T | T | |
|---|---|---|---|
| | | Serum Ferritin, % Transferrin Saturation) - Observed values, | |
| T | | Change and Percent Change from Baseline | T.A.G. |
| Table | Table 14.1.1.31 | Categorical Summary of Serum Ferritin, Serum Iron and % Transferrin Saturation | FAS |
| Table | | Serum Iron Indices (Total Iron Binding Capacity, Serum Iron, | FAS |
| | Table 14.1.1.32 | Serum Ferritin, % Transferrin Saturation) | |
| Table | | Serum Ferritin, Serum Total Iron, and % Transferrin | FAS |
| | | Saturation Values Meeting Categorical Summarization | |
| | Table 14.1.1.33 | Criteria | |
| Table | T 11 141 124 | Serum PF-06252616 Concentration (ng/mL) versus Time | FAS |
| T | Table 14.1.1.34 | Summary | T.A.G |
| Listing | Table 14.1.1.35 | Laboratory Abnormalities, by Cohort and Subject | FAS |
| Listing | Table 14.1.1.36 | Laboratory Abnormalities, by Dose Level and Subject | FAS |
| Listing | Table 14.1.1.37 | Laboratory Abnormalities, by Cohort, Dose Level and Test | FAS |
| | | Vital Signs | |
| Figure | Figure 14.1.1.1 | Vital Signs Absolute Values by Dose level | FAS |
| Figure | Figure 14.1.1.2 | Vital Signs Change from baseline by Dose Level | FAS |
| | | Electrocardiogram | |
| Table | Table 14.1.1.38 | Mean Baseline and Mean Changes from Baseline | FAS |
| Table | | Categorical Summary of Post-Baseline ECG Data - Absolute | FAS |
| | Table 14.1.1.39 | Values | |
| Table | | Categorical Summary of Post-Baseline ECG Data - Increases | FAS |
| | Table 14.1.1.40 | from Baseline | |
| Table | | Number (%) of Subjects with Single Uncorrected QT Values | FAS |
| | Table 14.1.1.41 | Greater than or Equal to 500 msec | |
| Table | Table 14.1.1.42 | ECG Change from Baseline | FAS |
| Table | Table 14.1.1.43 | ECG Qualitative Results | FAS |
| Table | T 11 14 1 1 44 | ECG Post-Baseline Values Meeting Categorical | FAS |
| E' | Table 14.1.1.44 | Summarization Criteria | EAG |
| Figure | | QTcF Interval (Fridericia's Correction) values over Time by | FAS |
| | F: 14112 | Dose Level - Box Plots | |
| Figure | Figure 14.1.1.3 | QTcF Interval (Fridericia's Correction) values change from | FAS |
| Figure | | , , | ras |
| | Figure 14.1.1.4 | baseline over Time by Dose Level - Box Plots | |
| Figure | Figure 14.1.1.4 | QT versus Heart Rate by Dose Level | FAS |
| rigure | Figure 14.1.1.5 | Q1 versus freatt Rate by Dose Level | TAS |
| | 1 iguic 14.1.1.5 | Cardiac MRI/Echocardiogram | |
| Table | | Shift Table of Left Ventricular Ejection Fraction over time by | FAS |
| Table | Table 14.1.1.45 | and Echocardiogram | I'AS |
| Table | 14010 1 1.1.1.13 | Mean absolute and percent change from baseline in Left | FAS |
| 10010 | Table 14.1.1.46 | Ventricular Ejection Fraction( LVEF) | |
| Table | | Mean absolute and percent change from baseline in Left | FAS |
| | Table 14.1.1.47 | Ventricular End Systolic Volume (LVESV) | |
| Listing | Table 14.1.1.48 | Echoardiagram | FAS |
| | | Liver MRI | |
| Table | | Summary of Average R2* Values and Percent Change from | FAS |
| | Table 14.1.1.49 | Baseline by Visit and Magnet Field Strength | |
| Table | Table 14.1.1.50 | Summary of Iron Accumulation | FAS |
| Table | Table 14.1.1.51 | Number (%) of Liver Enzyme Abnormalities by dose level | FAS |
| Listing | Table 14.1.1.52 | Liver Enzyme Abnormalities | FAS |
| Listing | Table 14.1.1.53 | Liver MRI | FAS |
| Listing | Table 14.1.1.54 | Liver MRI Abnormalities: R2* Elevations | FAS |

| | | DXA | FAS |
|---|---|---|---|
| Table | Table 14.1.1.55 | Bone Mineral Density over Time by Treatment (Whole Body) | FAS |
| Table | Table 14.1.1.56 | Bone Mineral Density over Time by Treatment (Hip) | FAS |
| Table | | Bone Mineral Density over Time by Treatment (Lumbar | FAS |
| | Table 14.1.1.57 | Spine) | |
| Listing | Table 14.1.1.58 | DXA | FAS |
| | | <b>Concomitant Medication</b> | |
| Listing | Table 14.1.1.59 | Concomitant Medications | FAS |
| | | CSSR | |
| Listing | Table 14.1.1.60 | C-SSRS by Time (Baseline/screen Version and Since last Visit) | FAS |
| Listing | Table 14.1.1.61 | C-SSRS by Time (Baseline/screen Version and Since last Visit) – Cont. | FAS |
| Table | Table 14.1.1.62 | | FAS |
| Table | 1 4010 14.1.1.02 | Anti-drug Antibodies (ADA) Status by Dose Level | TAS |
| Table | Table 14.1.1.62 | Secondary Endpoints: Summary of absolute value for Forced Vital Capcity (FVC) | EAC |
| Table Table | Table 14.1.1.63 Table 14.1.1.64 | Mean Change from Baseline for Forced Vital Capcity (FVC) | FAS |
| Table | 1 able 14.1.1.04 | Mean Forced Vital Capcity (FVC) | FAS<br>FAS |
| Table | | Mixed Model Repeated Measures (MMRM) of Change from | TAS |
| | Table 14.1.1.65 | Baseline | |
| Table | | Mean Forced Vital Capcity (FVC) | Completer Population |
| | | Mixed Model Repeated Measures (MMRM) of Change from | 1 1 |
| | Table 14.1.1.66 | Baseline | |
| Figure | Figure 14.1.1.6 | Plot of Mean Absolute Value on Frorced Vital Capcity | FAS |
| Figure | Figure 14.1.1.7 | Plot of Mean Change from Baseline on Frorced Vital Capcity | FAS |
| Table | Table 14.1.1.67 | Summary of absolute value for Performance of Upper Limb(PUL) | FAS |
| Table | | Mean Change from Baseline for Performance of Upper | FAS |
| T-1-1- | Table 14.1.1.68 | Limb(PUL) | FAS |
| Table | | Mean Performance of Upper Limb(PUL) Mixed Model Repeated Measures (MMRM) of Change from | FAS |
| | Table 14.1.1.69 | Baseline | |
| Table | 14010 14.1.1.09 | Mean Performance of Upper Limb(PUL) | Completer Population |
| Tuble | | Mixed Model Repeated Measures (MMRM) of Change from | Completer 1 optimion |
| | Table 14.1.1.70 | Baseline | |
| Table | Table 14.1.1.71 | Listing of Performance of Upper Limb | FAS |
| Listing | | Listing of items, Description and Scores Performance of | |
| | Table 14.1.1.72 | Upper Limb | |
| Figure | F: 14110 | Plot of Mean Absolute Value on Performance of Upper | FAS |
| E: | Figure 14.1.1.8 | Limb(PUL) | FAG |
| Figure | Figure 14.1.1.9 | Plot of Mean Change from Baseline on Performance of Upper Limb(PUL) | FAS |
| Table | Table 14.1.1.73 | Summary of absolute value for Timed Up & Go (TUG) | FAS |
| Table | Table 14.1.1.74 | Mean Change from Baseline for Timed Up & Go (TUG) | FAS |
| Table | 1 11.11.1 T | Mean Timed Up & Go (TUG) | FAS |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.75 | Baseline | |
| Table | | Mean Timed Up & Go (TUG) | Completer Population |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.76 | Baseline | |

| Figure | Figure 14.1.1.10 | Plot of Mean Absolute Value on Timed Up & Go (TUG) | FAS |
|---|---|---|---|
| Figure | <b>3</b> | Plot of Mean Change from Baseline on Timed Up & Go | FAS |
| 8 | Figure 14.1.1.11 | (TUG) | |
| Table | Table 14.1.1.77 | Summary of absolute value for for10-meter walk/run (10MR) | FAS |
| Table | Table 14.1.1.78 | Mean Change from Baseline for10-meter walk/run (10MR) | FAS |
| Table | | Mean 10-meter walk/run (10MR) | FAS |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.79 | Baseline | |
| Table | | Mean 10-meter walk/run (10MR) | Completer Population |
| | | Mixed Model Repeated Measures (MMRM) of Change from | 1 1 |
| | Table 14.1.1.80 | Baseline | |
| Figure | Figure 14.1.1.12 | Plot of Mean Absolute Value on 10-meter walk/run (10MR) | FAS |
| Figure | | Plot of Mean Change from Baseline on 10-meter walk/run | FAS |
| | Figure 14.1.1.13 | (10MR) | |
| Table | | Summary of absolute value for Two Minute Walk Test | FAS |
| | Table 14.1.1.81 | (2MWT) | |
| Table | | Mean Change from Baseline for Two Minute Walk Test | FAS |
| | Table 14.1.1.82 | (2MWT) | |
| Table | | Mean Two Minute Walk Test (2MWT) | FAS |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.83 | Baseline | |
| Table | | Mean Two Minute Walk Test (2MWT) | Completer Population |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.84 | Baseline | |
| Figure | 7 | Plot of Mean Absolute Value on Two Minute Walk Test | FAS |
| T. | Figure 14.1.1.14 | (2MWT)) | FAG |
| Figure | E: 14 1 1 15 | Plot of Mean Change from Baseline on Two Minute Walk | FAS |
| Table | Figure 14.1.1.15 Table 14.1.1.85 | Test (2MWT) Summary of absolute value for 4 Stair Climb (4SC) | FAS |
| Table | Table 14.1.1.86 | Mean Change from Baseline for 4 Stair Climb (4SC) | FAS |
| Table | 1 4016 14.1.1.60 | Mean 4 Stair Climb (4SC) | FAS |
| Table | | Mixed Model Repeated Measures (MMRM) of Change from | TAS |
| | Table 14.1.1.87 | Baseline | |
| Table | 14010 14.1.1.07 | Mean 4 Stair Climb (4SC) | Completer Population |
| Tubic | | Mixed Model Repeated Measures (MMRM) of Change from | Completel 1 optimion |
| | Table 14.1.1.88 | Baseline | |
| Figure | Figure 14.1.1.16 | Plot of Mean Absolute Value on 4 Stair Climb (4SC) | FAS |
| Figure | Figure 14.1.1.17 | Plot of Mean Change from Baseline on 4 Stair Climb (4SC) | FAS |
| Table | | Summary of absolute value for Forced Expiratory Volume in | FAS |
| | Table 14.1.1.89 | 1 second (FEV1) | |
| Table | | Mean Change from Baseline for Forced Expiratory Volume in | FAS |
| | Table 14.1.1.90 | 1 second (FEV1) | |
| Table | | Mean Forced Expiratory Volume in 1 second (FEV1) | FAS |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.91 | Baseline | |
| Table | | Mean Forced Expiratory Volume in 1 second (FEV1) | Completer Population |
| | m 11 - 11 - 1 | Mixed Model Repeated Measures (MMRM) of Change from | |
| - | Table 14.1.1.92 | Baseline | 7.40 |
| Figure | TO: 144.440 | Plot of Mean Absolute Value on Forced Expiratory Volume | FAS |
| T71 | Figure 14.1.1.18 | in 1 second (FEV1) | FAG |
| Figure | E' 141110 | Plot of Mean Change from Baseline on Forced Expiratory | FAS |
| T. 11 | Figure 14.1.1.19 | Volume in 1 second (FEV1) | EAC |
| Table | Table 14 1 1 02 | Summary of absolute value for Maximal Inspiratory Pressure | FAS |
| Table | Table 14.1.1.93 | (MIP) Mean Change from Passline for Maximal Inchiratory | EAC |
| Table | Table 14.1.1.94 | Mean Change from Baseline for Maximal Inspiratory | FAS |

| | | Pressure (MIP) | |
|---|---|---|---|
| Table | | Mean Maximal Inspiratory Pressure (MIP) | FAS |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.95 | Baseline | |
| Table | | Mean Maximal Inspiratory Pressure (MIP) | FAS |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.96 | Baseline | |
| Figure | | Plot of Mean Absolute Value on Maximal Inspiratory | FAS |
| | Figure 14.1.1.20 | Pressure (MIP) | |
| Figure | F: 141101 | Plot of Mean Change from Baseline on Maximal Inspiratory | FAS |
| T 11 | Figure 14.1.1.21 | Pressure (MIP) | T.A.C. |
| Table | T-1-1-141107 | Summary of absolute value for Maximal Expiratory Pressure | FAS |
| Table | Table 14.1.1.97 | (MEP) | FAS |
| Table | Table 14 1 1 09 | Mean Change from Baseline for Maximal Expiratory Pressure (MEP) | ras |
| Table | Table 14.1.1.98 | Mean Maximal Expiratory Pressure (MEP) | FAS |
| Table | | Mixed Model Repeated Measures (MMRM) of Change from | ras |
| | Table 14.1.1.99 | Baseline | |
| Table | 14010 1 1.11.11.99 | Mean Maximal Expiratory Pressure (MEP) | Completer Population |
| 1 4010 | | Mixed Model Repeated Measures (MMRM) of Change from | Completer reputation |
| | Table 14.1.1.100 | Baseline | |
| Figure | Figure 14.1.1.22 | Plot of Mean Absolute Value on Expiratory Pressure (MEP) | FAS |
| Figure | | Plot of Mean Change from Baseline on Maximal Expiratory | FAS |
| | Figure 14.1.1.23 | Pressure (MEP) | |
| Table | | Summary of absolute value for Muscle Strength BY Manual | FAS |
| | Table 14.1.1.101 | Muscle Test (MMT) and Hand-Hels dynamometry | |
| Table | | Mean Change from Baseline for Muscle Strength BY Manual | FAS |
| | Table 14.1.1.102 | Muscle Test (MMT) and Hand-Hels dynamometry | |
| Table | | Mean Muscle Strength BY Manual Muscle Test (MMT) and | FAS |
| | | Hand-Hels dynamometry | |
| | Table 14.1.1.103 | Mixed Model Repeated Measures (MMRM) of Change from Baseline | |
| Table | 1 4.1.1.103 | Mean Muscle Strength BY Manual Muscle Test (MMT) and | Completer Population |
| Table | | Hand-Hels dynamometry | Completed Topulation |
| | | Mixed Model Repeated Measures (MMRM) of Change from | |
| | Table 14.1.1.104 | Baseline | |
| Listing | | Listing of Manual Muscle Test (MMT) and Hand-Helded | FAS |
| C | Table 14.1.1.105 | dynamometry (Manual Muscle Test) | |
| Listing | | Listing of Manual Muscle Test (MMT) and Hand-Helded | FAS |
| | Table 14.1.1.106 | dynamometry (Hand Held Myometry) | |
| Figure | | Plot of Mean Absolute Value on Muscle Strength BY Manual | FAS |
| | Figure 14.1.1.24 | Muscle Test (MMT) and Hand-Hels dynamometry | |
| Figure | | Plot of Mean Change from Baseline on Muscle Strength BY | FAS |
| | Figure 14.1.1.25 | Manual Muscle Test (MMT) and Hand-Hels dynamometry | |
| Table | Table 14.1.1.107 | Total Score for InQol | FAS |
| Table | Table 14.1.1.108 | InQol: Summary Statistics for Weakness Symptom | FAS |
| Table | Table 14.1.1.109 | InQol: Summary Statistics for Locking Symptom FAS | |
| Table | Table 14.1.1.110 | | |
| Table | Table 14.1.1.111 | | |
| Table | Toble 14 1 1 112 | SF-36 Questionnaire: Listing of Physical and Mental FAS | |
| | Table 14.1.1.112 | CDE 9 Concentration | |
| Table | | GDF-8 Concentration Sarum Total GDF 8 Concentration (NG/ML) warsus Time | |
| rabie | Table 14.1.1.113 | Serum Total GDF-8 Concentration (NG/ML) versus Time Listing | |
| | 1 4010 17.1.1.113 | Listing | 1 |

| | I | THE THE THE THE PERSON OF THE |
|---|---|---|
| Figure | | Individual Serum Total GDF-8 Concentration (NG/ML) - |
| | Figure 14.1.1.25 | Time Plot by Cohort (Linear Scale) |
| Figure | | Individual Change from Baseline of Serum Total GDF-8 |
| | Figure 14.1.1.26 | Concentration (NG/ML) - Time Plot by Cohort (Linear Scale) |
| Table | Table 14.1.1.114 | Serum Total GDF-8 (NG/ML) versus Time Summary |
| Table | Table 14.1.1.115 | Changes from Baseline for Serum Total GDF-8 (NG/ML) |
| Figure | | Median Serum Total GDF-8 Concentration (NG/ML) - Time |
| | Figure 14.1.1.27 | Plot by Cohort (Linear Scale) |
| Figure | | Median Change from Baseline of Serum Total GDF-8 |
| | Figure 14.1.1.28 | Concentration (NG/ML) - Time Plot by Cohort (Linear Scale) |
| Figure | | Mean Serum Total GDF-8 Concentration (NG/ML) - Time |
| | Figure 14.1.1.29 | Plot by Cohort (Linear Scale) |
| Figure | | Mean Change from Baseline of Serum Total GDF-8 |
| | Figure 14.1.1.30 | Concentration (NG/ML) - Time Plot by Cohort (Linear Scale) |
| Figure | | Median Serum Total GDF-8 Concentration (NG/ML) - Time |
| | Figure 14.1.1.31 | Plot by Cohort (Linear Scale) |
| Figure | | Median Change from Baseline of Serum Total GDF-8 |
| 8 | Figure 14.1.1.32 | Concentration (NG/ML) - Time Plot by Cohort (Linear Scale) |
| Figure | Table 14.1.1.116 | Descriptive Summary of Serum Total GDF-8 Parameters |
| | | PK Summary |
| Table | | Serum PF-06252616 Concentration [NG/MG] versus Time |
| | Table 14.1.1.117 | Summary for All Subjects |
| Table | | Serum PF-06252616 Concentration [NG/MG] versus Time |
| | Table 14.1.1.118 | Summary for Subjects with Additional Sampling |
| Figure | | Median Serum PF-06252616 Concentration - Time Plot by |
| | Figure 14.1.1.33 | Cohort (Linear Scale) for All Subjects |
| Figure | <u> </u> | Median Serum PF-06252616 Concentration - Time Plot by |
| | Figure 14.1.1.34 | Cohort (Linear Scale) for Subjects with Additional Sampling |
| Figure | | Mean Serum PF-06252616 Concentration - Time Plot by |
| | Figure 14.1.1.35 | Cohort (Linear Scale) for All Subjects |
| Figure | | Mean Serum PF-06252616 Concentration - Time Plot by |
| | Figure 14.1.1.36 | Cohort (Linear Scale) for Subjects with Additional Sampling |
| Figure | | Median Serum PF-06252616 Concentration - Time Plot by |
| | Figure 14.1.1.37 | Cohort (Linear Scale) for All Subjects |
| Figure | _ | Median Trough Serum PF-06252616 Concentration - Time |
| | Figure 14.1.1.38 | Plot by Cohort (Linear Scale) |
| Figure | _ | Median End of Infusion Serum PF-06252616 Concentration - |
| | Figure 14.1.1.39 | Time Plot by Cohort (Linear Scale) |
| Table | _ | Descriptive Summary of Serum PF-06252616 PK Parameters |
| | Table 14.1.1.119 | for All Subjects |
| Table | | Descriptive Summary of Serum PF-06252616 PK Parameters |
| | Table 14.1.1.120 | for Subjects with Additional PK Sampling |
| Table | | Descriptive Summary of Serum PF-06252616 PK Parameters |
| | Table 14.1.1.121 | for All Subjects – Process 1 vs Process 2 |
| | • | |



# CLINICAL AND MEDICAL CONTROLLED DOCUMENT (CMCD) REQUIRED FORM

| Identifier | Version | Title | Effective Date |
|---|---|---|---|
| DMB02-GSOP-<br>RF01 | 6.0 | STATISTICAL ANALYSIS PLAN<br>APPROVAL SIGNATURE FORM | 01-Nov-2018 |

**NOTE:** This form is used to document the approval of a Statistical Analysis Plan (SAP) and any subsequent amendment of the SAP.

| SAP Title: Include protocol number and format per following example: A### Statistical Analysis Plan | AWI203720 Statistical Analysis Plan |
|---|---|
| Approval of SAP Approval of Amendment to SAP | SAP Version: 1.0 |

| Name and Title of Person Submitting form: (SAP Author) | Nazila Shahri |
|--------------------------------------------------------|---------------|
| | 12 Feb 2019 |

Approval indicates that the SAP provides analysis specifications consistent with the analysis outlined in the protocol and meets the standards and requirements used for programming of tables, listings and figures.

| igures. | |
|--------------------------|-----------------------------------------|
| SAP Approver's<br>Name: | Nazila Shahri |
| SAP Approver's<br>Title: | Statistician |
| Signature: | NI. Shahri |
| (dd-Mmm-yyyy) | 12 Feb 2019 |
| SAP Approver's<br>Name: | Jeffrey Palmer |
| SAP Approver's<br>Title: | Senior Director, Biostatistics (Pfizer) |

| Signature: | | |
|--------------------------------|-------------------------|---|
| <b>Date:</b><br>(dd-Mmm-yyyy) | 12-FEB-2019 | |
| SAP Approver's<br>Name: | Kathryn Wagner | |
| SAP Approver's<br>Title: | Principal Investigator | |
| Signature: | algrer | |
| Date:<br>(dd-Mmm-yyyy) | 12 FEB Zaig | |
| SAP Approver's<br>Name: | Shirley Galbiati | |
| SAP Approver's<br>Title: | Biostatistician (Emmes) | |
| Signature: | Shelah | • |
| Da <b>ţe:</b><br>(dd-Mmm-yyyy) | 12 Feb 2019. | |